CLINICAL TRIAL: NCT07051187
Title: An Open-Label, Single-Arm, Dose-Escalation Phase I Clinical Trial to Evaluate the Efficacy and Safety of WGc0201 in Patients With Chronic Hepatitis B Virus Infection
Brief Title: A Trial to Evaluate the Efficacy and Safety of WGc0201 in Patients With Chronic Hepatitis B Virus Infection
Acronym: WGc0201-HBV
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiyan Liu (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor-Investigator, Jiyan Liu, Deputy Director of the Department of Biotherapy, West China Hospital, Sichuan University, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WGc0201-HBV-001; 274953 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2025-05-30; First posted 2025-07-04 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hepatitis B Virus (Hbv)
Keywords: mRNA; vaccine; chronic Hepatitis B virus
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WGc0201 (Experimental): Wgc0201 will be administered by intramuscular route, with a total of 9 doses
  Interventions: Drug: WGc0201

INTERVENTIONS:
Drug: WGc0201 — Wgc0201 will be administered by intramuscular route, with a total of 9 doses.

SUMMARY:
Existing nucleoside analogues (NAs) and interferon therapy for chronic hepatitis B (CHB) have limitations, including drug resistance, low HBsAg clearance rates, and irreversible immunosuppression. Therapeutic vaccines, by activating virus-specific T cells and B cells, hold promise for achieving functional cure (HBsAg clearance + sustained HBV DNA negativity). This study is an open-label, single-arm, dose-escalation Phase I clinical trial. The study population consists of patients with chronic hepatitis B virus infection who have achieved virological stability following standard antiviral therapy. Phase I (dose exploration): three dose groups, with three patients per group. The primary objective is to observe and evaluate the safety of the WGc0201 vaccine in the study population (incidence and severity of adverse events).

DETAILED DESCRIPTION:
Although current antiviral treatments have achieved some clinical efficacy, there is still a lack of treatments that can truly cure hepatitis B, especially those that can completely eliminate HBsAg and prevent viral recurrence. Therapeutic hepatitis B vaccines are considered a potential treatment option for chronic hepatitis B and drug-resistant hepatitis B patients in the future. The development goal of therapeutic vaccines is to activate the body's specific immune response, promote the immune system to recognize and eliminate the hepatitis B virus, thereby achieving virological clearance and functional cure. WGc-0201 injection is an mRNA vaccine encoding the HBV-positive tumor antigen HBx. Preliminary basic research conducted by the team suggests that this vaccine has excellent safety, not only effectively clearing HBV DNA but also reducing HBsAg levels in serum and liver tissue while enhancing the expansion of specific T lymphocytes in the body. Therefore, we believe that the efficacy and safety of WGc0201 in treating hepatitis B warrant further investigation. We aim to use this Phase I study to preliminarily explore the therapeutic efficacy and safety of WGc0201 in this population and lay the groundwork for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females aged ≥18 to ≤65 years;
2. 18≤ BMI ≤32 kg/m2;
3. Diagnosis of chronic hepatitis B infection (HBsAg positive for more than 6 months and detectable at screening);
4. Received only nucleoside (acid) analog therapy in the 12 months prior to screening and are still taking it regularly;
5. HBV-DNA viral load below 100 IU/ml;
6. HBsAg <1500 IU/ml.

Exclusion Criteria:

1. Includes HIV, co-infection with HDV, and liver biopsy suggestive of cirrhosis or advanced fibrosis within 6 months prior to screening (Metavir activity level A3 and stages F3 and F4; Ishak stages 4-6);
2. If no liver biopsy was documented, a Fibroscan screen result >9 kPa (or equivalent) or a FibroTest screen result >0.48 and an APRI (Aspartate Aminotransferase to Platelet Ratio Index) >1 within ≤6 months of screening.
3. Alanine aminotransferase >3x ULN;
4. Internationally standardized ratio > 1.5;
5. Albumin <3.5 g/dl;
6. Direct bilirubin > 1.5x ULN;
7. Platelet count <100,000/μl;
8. History of hepatic failure (e.g., ascites, encephalopathy, or variceal bleeding) or prior hepatocellular carcinoma;
9. Diseases or past history of the following systems or serious illnesses that the investigator considers inappropriate for participation in this trial, such as: cardiovascular system: unstable or significant cardiovascular disease, such as angina pectoris, recent episode of myocardial infarction, congestive heart failure, severe hypertension, significant arrhythmia or ECG abnormality, etc.; respiratory system: bronchiectasis, bronchial asthma, chronic obstructive pulmonary disease, respiratory failure, etc.; endocrine and metabolic diseases: diabetes mellitus, thyroid disease poorly controlled by medication, etc.; others: autoimmune diseases, active tuberculosis, malignant diseases (e.g., tumors), history of neurological or psychiatric disorders, etc;
10. Subjects who have participated in any drug/device clinical study within 3 months prior to receiving the experimental drug.
11. History of organ transplantation (except corneal transplantation and hair transplantation).
12. Those with alcoholism (alcohol consumption for more than 5 years prior to the screening period, with alcohol content greater than 40g per day for men and 20g per day for women) or known drug dependence.
13. Subjects who have a birth plan or a plan to donate sperm or eggs during the screening period, during the trial, and for 6 months after the end of the trial or who are unwilling to use effective contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | 12 weeks
  CATAE 5.0 standard

SECONDARY OUTCOMES:
Immunogenicity of the vaccine (HBV-specific T-cell response) | 12 weeks
  ELISpot test
changes in virological indicators (HBV DNA/RNA) | 12 weeks
  qPCR、RT-qPCR
changes in virological indicators (HBsAg) | 12 weeks
  CLIA/ECLIA
changes in virological indicators (ALT normalization rate) | 12 weeks
  Kinetic (Rate) Assay

IPD SHARING:
Plan to Share IPD: No